CLINICAL TRIAL: NCT01485198
Title: Clinical Effects of Autologous Bone Marrow Mononuclear Cell Infusion in Knee Osteoarthritis.
Brief Title: Autologous Stem Cells in Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Consuelo Mancias Guerra, Head of Hematology Service, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE11-022
Record Dates: First submitted 2011-11-26; First posted 2011-12-05 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; stem cell therapy; bone marrow; G-CSF
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Patients treated with Acetaminophen
  Interventions: Drug: Acetaminophen
- Experimental (Experimental): Patients who underwent a BMASC extraction and joint infusion
  Interventions: Procedure: Bone Marrow Autologous Stem Cells Infusion

INTERVENTIONS:
Procedure: Bone Marrow Autologous Stem Cells Infusion — Extraction and knee infusion of Bone Marrow Autologous Stem Cells
  Other Names: Knee treatment with stem cells
  Arms: Experimental
Drug: Acetaminophen — Acetaminophen (750mg orally TID) administration
  Other Names: Knee treatment with NSAIDs
  Arms: Control

SUMMARY:
Patients with osteoarthritis, a degenerative joint disease, that meet inclusion criteria will be allocated into two groups:

* The control group will receive Acetaminophen 750mg orally every 8 hours
* The experimental group will receive Autologous Hematopoietic Stem Cells from bone marrow (BMASC)

Signed informed consent is required, as well as answering a questionnaire.

Patients in experimental group will receive subcutaneous G-CSF (10ug/kg/day) for 3 consecutive days and, on the 4th day a bone marrow harvest under general sedation will be performed from posterior iliac crests. The patient will remain in the recovery room while the cells are processed at the Hematology Service Laboratory. Finally, BMASC will be infused to the joint under local anesthesia.

The procedure is ambulatory.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee osteoarthritis grade II or III of the Kellgren-Lawrence radiographic scale
* Age > 30 years

Exclusion Criteria:

* Neurodegenerative, autoimmune, genetic or psychiatric diseases
* Active infection
* Recent joint infection
* Knee surgery history
* Knee joint fracture history

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Define safety of BM extraction and stem cell joint infusion. | 1 week
  Measure possible complications of procedure (e.g. pain, bleeding, infection) and range of motion through clinical examination.
  Apply a questionnaire consisting of validated Womac® Scale, KSS® (Knee Society Rating System), SF-36® (Health Survey Update), and VAS (Visual Analog Scale) to correlate changes at first week to the baseline questionnaire.

SECONDARY OUTCOMES:
Efficacy of BMSC joint infusion at 4 weeks | 4 weeks
  Measure possible complications of procedure (e.g. pain, bleeding, infection) and range of motion through clinical examination.
  Apply a questionnaire consisting of validated Womac® Scale, KSS® (Knee Society Rating System), SF-36® (Health Survey Update), and VAS (Visual Analog Scale) to correlate changes with first week and baseline questionnaires.
Efficacy and final outcome of BMSC joint infusion at 6 months. | 24 weeks
  Measure possible complications of procedure (e.g. pain, bleeding, infection) and range of motion through clinical examination.
  Apply a questionnaire consisting of validated Womac® Scale, KSS® (Knee Society Rating System), SF-36® (Health Survey Update), and VAS (Visual Analog Scale) to correlate changes with 4 week, first week and baseline questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Domingo Garay Mendoza, MD, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez; Consuelo Mancias Guerra, MD, Study Director — Hospital Universitario Dr. Jose E. Gonzalez; Laura Villarreal Martínez, MD, Study Chair — Hospital Universitario Dr. Jose E. Gonzalez
Locations (2):
- Mexico (2):
  - Hematology Service, Monerrey, Nuevo León
  - Traumatology Service, Monterrey, Nuevo León

REFERENCES:
- [Result] Davatchi F, Abdollahi BS, Mohyeddin M, Shahram F, Nikbin B. Mesenchymal stem cell therapy for knee osteoarthritis. Preliminary report of four patients. Int J Rheum Dis. 2011 May;14(2):211-5. doi: 10.1111/j.1756-185X.2011.01599.x. Epub 2011 Mar 4. PMID 21518322
- [Result] de Girolamo L, Bertolini G, Cervellin M, Sozzi G, Volpi P. Treatment of chondral defects of the knee with one step matrix-assisted technique enhanced by autologous concentrated bone marrow: in vitro characterisation of mesenchymal stem cells from iliac crest and subchondral bone. Injury. 2010 Nov;41(11):1172-7. doi: 10.1016/j.injury.2010.09.027. Epub 2010 Oct 8. PMID 20934693
- [Result] Chen FM, Wu LA, Zhang M, Zhang R, Sun HH. Homing of endogenous stem/progenitor cells for in situ tissue regeneration: Promises, strategies, and translational perspectives. Biomaterials. 2011 Apr;32(12):3189-209. doi: 10.1016/j.biomaterials.2010.12.032. PMID 21300401
- [Derived] Garay-Mendoza D, Villarreal-Martinez L, Garza-Bedolla A, Perez-Garza DM, Acosta-Olivo C, Vilchez-Cavazos F, Diaz-Hutchinson C, Gomez-Almaguer D, Jaime-Perez JC, Mancias-Guerra C. The effect of intra-articular injection of autologous bone marrow stem cells on pain and knee function in patients with osteoarthritis. Int J Rheum Dis. 2018 Jan;21(1):140-147. doi: 10.1111/1756-185X.13139. Epub 2017 Jul 27. PMID 28752679
- See also: Traumatology Service Web Site — http://www.ortopedia.org/